CLINICAL TRIAL: NCT01482845
Title: A Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ABT-126 in Subjects With Alzheimer's Disease on Stable Doses of Acetylcholinesterase Inhibitors
Brief Title: A Phase 1 Study of the Safety, Tolerability and Pharmacokinetics of ABT-126 in Subjects With Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: M12-970
Record Dates: First submitted 2011-11-21; First posted 2011-12-01 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-03

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — ABT-126

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental)
  Interventions: Drug: ABT-126; Drug: Placebo
- Group 2 (Experimental)
  Interventions: Drug: ABT-126; Drug: Placebo

INTERVENTIONS:
Drug: ABT-126 — Dose 1 is given to 8 subjects in Group 1. Dose 2 is given to 8 subjects in Group 2. All doses will be administered once daily in the morning for 10 days.
Drug: Placebo — Placebo is given to 2 subjects each in Group 1 and Group 2. All doses will be administered once daily in the morning for 10 days.

SUMMARY:
This study will investigate safety, tolerability and pharmacokinetics of ABT-126 in up to 20 male and female subjects, between 55 to 90 years of age with mild to moderate Alzheimer's disease on stable doses of acetylcholinesterase inhibitors.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, randomized, multiple-dose, parallel group, multicenter study. Up to 20 male and female subjects with mild to moderate Alzheimer's disease (AD) who are taking stable doses of acetylcholinesterase inhibitors will be enrolled in this study. The study will be conducted in up to four sites. Within 28 days prior to study drug administration, subjects will be screened based on National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria for probable AD, Mini-Mental State Examination (MMSE) and Modified Hachinski Ischemic Scale (MHIS) scores, medical history, physical examination, neurological examination, vital signs, ECG, laboratory tests and response to Columbia-Suicide Severity Rating Scale (C-SSRS).

Subjects will be divided into two groups of 10 subjects each. In each group, 8 subjects will receive ABT-126 and two subjects will receive matching placebo. Group 1 will be administered Dose 1 of ABT-126 or placebo. Group 2 will be administered Dose 2 ABT-126 or placebo. All doses will be administered once daily in the morning for 10 days.

ELIGIBILITY:
Inclusion Criteria

1. Male or female and age between 55 and 90 years, inclusive.
2. The subject meets the National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria for probable Alzheimer's Disease (AD).
3. The subject has a Mini-Mental State Examination (MMSE) total score of 16 to 26, inclusive, at Screening Visit.
4. The subject has a Modified Hachinski Ischemic Scale (MHIS) score of ≤ 4 at Screening Visit.
5. The subject must be on a stable dose of donepezil or rivastigmine for at least 1 month prior to study drug administration.
6. The subject has had a computerized tomography or magnetic resonance imaging scan, interpreted by a radiologist or neurologist, within 36 months prior to randomization and after the subject met NINCDS/ADRDA diagnostic criteria for probable AD. The scan must not show evidence for an alternative etiology for dementia.

Exclusion Criteria

1. Receipt of an investigational product within 6 weeks prior to study drug administration.
2. History of significant sensitivity or allergy to any drug.
3. History of any significant neurological disease other than AD.
4. Significant current suicidal ideation within 1 month prior to study drug administration as evidenced by answering "yes" to questions 4 or 5 on the suicidal ideation portion of the Columbia-Suicide Severity Rating Scale (C-SSRS) completed at Screening or any history of suicide attempts.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessments | From Day 1 through Day 17
  vital signs, electrocardiogram (ECG), neurological examination, laboratory tests, number of subjects with adverse events, Columbia-Suicide Severity Rating Scale (C-SSRS)

SECONDARY OUTCOMES:
Pharmacokinetic evaluation profile | Blood collection prior to, and at 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24, 72, 120, and 168 hours after dosing on Day 10
  Area under curve (AUC), maximum concentration(Cmax), minimum concetration (Cmin), time to peak concentration (Tmax), half-life(t1/2), clearance (CL/F)

CONTACTS AND LOCATIONS:
Overall Officials: Hana Florian, MD, Study Director — Abbott
Locations (3):
- United States (3):
  - Site Reference ID/Investigator# 62908, Glendale, California
  - Site Reference ID/Investigator# 62904, Hallandale, Florida
  - Site Reference ID/Investigator# 62903, Orlando, Florida